CLINICAL TRIAL: NCT03270267
Title: Chronic Inflammatory Bowel Diseases and School Absenteeism
Brief Title: Chronic Inflammatory Bowel Diseases (IBD) and School Absenteeism
Acronym: MICI School
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3035_MICI School
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with IBD
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires

SUMMARY:
Study of the causes and rate of school absenteeism in children and adolescents with Inflammatory Bowel Disease.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6 to 18 years old
* Child with definite diagnosis of IBD for at least 6 months
* Follow-up by a gastroenterologist of Rennes University Hospital on a regular basis (at least 2 annual consultations)
* Non-opposition of the child and the parents

Exclusion Criteria:

* School leaving
* Student at the University
* Other serious disease outside IBD preventing normal schooling
* Refusal of participation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with IBD
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Number of days of absence from school due to IBD | Month 10

SECONDARY OUTCOMES:
Comparison of the rate of school absenteeism of a child with IBD to the data of the school academy where she/he is enrolled | Month 10
Study of repercussion of the number of days of absence due to IBD on school results | Month 10

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France